CLINICAL TRIAL: NCT07221708
Title: Primary Prophylaxis of Clostridioides Difficile Infection With Oral Vancomycin in Patients Treated With Systemic Antibiotic Therapy in a Community Hospital
Brief Title: Primary Prophylaxis of Clostridioides Difficile Infection With Oral Vancomycin
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: University of Maryland, Baltimore Washington Medical Center (Unknown)
Responsible Party: Principal Investigator, Jeffrey Marshall, Associate Chief Medical Officer and VP of Quality and Patient Safety, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HP-00113868
Record Dates: First submitted 2025-10-17; First posted 2025-10-28 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Clostridioides Difficile; Vancomycin Resistance Enterococcus Faecium
Keywords: Clostridioides Difficile; Vancomycin Resistance Enterococcus faecium; C Diff; VRE; Vancomycin; C Diff Infection
MeSH Terms: conditions — Clostridium Infections | interventions — Vancomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral Vancomycin (Experimental): The oral vancomycin treatment group will receive oral vancomycin 125 mg twice daily for the duration of the concomitant antibiotic plus two additional days.
  Interventions: Drug: Vancomycin (POC)
- No Oral Vancomycin (No Intervention): The no oral vancomycin control group will receive the current standard of care treatment which is an antibiotic with no oral vancomycin.

INTERVENTIONS:
Drug: Vancomycin (POC) — A dosage of oral vancomycin 125 mg will be given twice daily for the duration of the concomitant antibiotic plus two additional days
  Arms: Oral Vancomycin

SUMMARY:
The purpose of this study is to evaluate the ability of oral vancomycin in preventing Clostridioides difficile infection (CDI) in patients that are simultaneously receiving antibiotics.

Participants in this study will be placed randomly into two groups. The oral vancomycin treatment group will receive oral vancomycin two times per day simultaneously with an antibiotic plus two additional days. The no oral vancomycin control group will receive the current standard of care, which is an antibiotic and no oral vancomycin. Participation in this study will last approximately 3 months.

DETAILED DESCRIPTION:
This research study is being conducted to evaluate the feasibility of prescribing oral vancomycin in preventing CDI in patients who are receiving concomitant systemic antibiotics.

There are two groups: one group will receive oral vancomycin 125 mg twice daily for the duration of systemic antibiotic use plus two additional days; the other group will receive the current standard of care which is no oral vancomycin. The investigators aim to collect data from 100 patients in each group for a total of 200 patients.

Eligible participants will be randomized in a 1:1 ratio to receive either oral vancomycin or no oral vancomycin. A computer-generated randomization sequence has been created using block randomization with variable block sizes (4, 6, 8) to maintain group balance and reduce predictability.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years or older
* Receive systemic antibiotics in the last 90 days
* Hospitalized anywhere in the last 90 days
* History of C diff colonization without history of C diff colitis (infection)
* Provide informed consent
* Read and understand the English language
* Not current taking probiotics
* Lack of allergy or contraindications to receive vancomycin
* Ability to take oral medications
* Not receiving medications that can be used to treat or prevent C diff

Exclusion Criteria:

* Age 64 years or younger
* Has not received systemic antibiotics in the last 90 days
* Has not been hospitalized in the last 90 days
* History of C diff colonization with a history of C diff colitis (infection)
* Not provided informed consent
* Cannot read and understand the English language
* Currently receiving probiotics
* Allergy or contraindications to receive vancomycin
* Unable to take oral medications
* Receiving medications that can be used to treat or prevent C diff

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants who develop C diff after receiving oral vancomycin plus another antibiotic at the same time versus participants who do not receive oral vancomycin | Hospitalization duration and through 90 days post hospitalization discharge

SECONDARY OUTCOMES:
Number of participants who develop vancomycin resistant enterococcus | At start of study participation (baseline) and at completion of antibiotics (up to four weeks).
  Perirectal swabs to detect vancomycin-resistant Enterococcus (VRE) will be performed at the time of study inclusion and repeated at discharge. The investigators will use this data to evaluate acquisition of resistance following exposure to vancomycin.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Marshall, MD, Principal Investigator — University of Maryland, Baltimore Washington Medical Center
Locations (1):
- University of Maryland Baltimore Washington Medical Center, Glen Burnie, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ganetsky A, Han JH, Hughes ME, Babushok DV, Frey NV, Gill SI, Hexner EO, Loren AW, Luger SM, Mangan JK, Martin ME, Smith J, Freyer CW, Gilmar C, Schuster M, Stadtmauer EA, Porter DL. Oral Vancomycin Prophylaxis Is Highly Effective in Preventing Clostridium difficile Infection in Allogeneic Hematopoietic Cell Transplant Recipients. Clin Infect Dis. 2019 May 30;68(12):2003-2009. doi: 10.1093/cid/ciy822. PMID 30256954
- [Background] Papic N, Maric LS, Vince A. Efficacy of oral vancomycin in primary prevention of Clostridium Difficile infection in elderly patients treated with systemic antibiotic therapy. Infect Dis (Lond). 2018 Jun;50(6):483-486. doi: 10.1080/23744235.2018.1425551. Epub 2018 Jan 11. No abstract available. PMID 29323607
- [Background] Maraolo AE, Mazzitelli M, Zappulo E, Scotto R, Granata G, Andini R, Durante-Mangoni E, Petrosillo N, Gentile I. Oral Vancomycin Prophylaxis for Primary and Secondary Prevention of Clostridioides difficile Infection in Patients Treated with Systemic Antibiotic Therapy: A Systematic Review, Meta-Analysis and Trial Sequential Analysis. Antibiotics (Basel). 2022 Jan 30;11(2):183. doi: 10.3390/antibiotics11020183. PMID 35203786
- [Background] Tariq R, Laguio-Vila M, Tahir MW, Orenstein R, Pardi DS, Khanna S. Efficacy of oral vancomycin prophylaxis for prevention of Clostridioides difficile infection: a systematic review and meta-analysis. Therap Adv Gastroenterol. 2021 Feb 23;14:1756284821994046. doi: 10.1177/1756284821994046. eCollection 2021. PMID 33747124
- [Background] Johnson SW, Brown SV, Priest DH. Effectiveness of Oral Vancomycin for Prevention of Healthcare Facility-Onset Clostridioides difficile Infection in Targeted Patients During Systemic Antibiotic Exposure. Clin Infect Dis. 2020 Aug 22;71(5):1133-1139. doi: 10.1093/cid/ciz966. PMID 31560051